CLINICAL TRIAL: NCT01991665
Title: Randomised Italian Sonography for Occiput POSition Trial Ante Vacuum
Brief Title: R. I. S. POS. T. A
Acronym: RISPOSTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Tullio Ghi, Dr T. Ghi, Obstetrics and Prenatal Medicine Unit, University Hospital of Parma, University of Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OST-2013-50
Record Dates: First submitted 2013-11-17; First posted 2013-11-25 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Vacuum Extraction; Failure, Affecting Fetus or Newborn; Persistent Occiput Posterior Position During Labor; Complication of Delivery
Keywords: Intrapartum Ultrasound; Vacuum; Occiput position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): Digital examination before instrumental delivery to determine fetal head station and position
  Interventions: Other: Digital examination
- Group B (Other): Digital examination before instrumental delivery to determine fetal head station and position + sonography evaluation of fetal head position
  Interventions: Other: Digital examination; Other: Sonography evaluation

INTERVENTIONS:
Other: Digital examination
Other: Sonography evaluation
  Arms: Group B

SUMMARY:
A failed operative vaginal delivery is associated with increased risk of maternal and perinatal complications. It is very important the determination of the fetal head position prior to instrumental delivery.

Generally,diagnosis of the fetal head position is made on transvaginal digital examination by delineating the suture lines of the fetal skull and the fontanelles. There is a paucity of studies on the accuracy of digital examination but the general consensus is that reproducibility is low and diagnostic uncertainty remains high even for operators with much experience.

As the traditional clinical evaluation has many limitations, a new tool capable of increasing diagnostic objectivity and accuracy would be of great interest.

The aim of our study was to evaluate, in a prospective study, if the complementary use of ultrasound scan, to diagnose the fetal head position prior to instrumental delivery, may play a role in labor outcome.

ELIGIBILITY:
Inclusion Criteria:

* women with singleton cephalic pregnancies at term (≥37 weeks' gestation), who require an instrumental delivery

Exclusion Criteria:

* under 18 years of age
* women with contraindications for vacuum delivery
* women with sonography evaluation of fetal head position before randomization
* fetal head station > +3
* discretion of the responsible obstetrician in cases where there is urgency due to suspected fetal compromise("fetal distress")

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1400 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
failure rate of vacuum extraction in each of the two groups of patients included in the study (number of cesarean deliveries). | 2 years

SECONDARY OUTCOMES:
Incidence of: neonatal trauma (cephalhaematoma, retinal haemorrhage, facial nerve palsy, brachial plexus injury and fractures), low Apgar scores, fetal acidosis or admission to the neonatal unit, shoulder dystocia | 2 years
Incidence of: primary postpartum haemorrhage, third and fourth degree perineal tears | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tullio Ghi, Principal Investigator — Department of Obstetrics and Gynecology, Sant'Orsola-Malpighi Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Sant'Orsola-Malpighi University Hospital, University of Bologna, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Background] Groutz A, Hasson J, Wengier A, Gold R, Skornick-Rapaport A, Lessing JB, Gordon D. Third- and fourth-degree perineal tears: prevalence and risk factors in the third millennium. Am J Obstet Gynecol. 2011 Apr;204(4):347.e1-4. doi: 10.1016/j.ajog.2010.11.019. Epub 2010 Dec 22. PMID 21183150
- [Background] Towner D, Castro MA, Eby-Wilkens E, Gilbert WM. Effect of mode of delivery in nulliparous women on neonatal intracranial injury. N Engl J Med. 1999 Dec 2;341(23):1709-14. doi: 10.1056/NEJM199912023412301. PMID 10580069
- [Background] Dupuis O, Silveira R, Zentner A, Dittmar A, Gaucherand P, Cucherat M, Redarce T, Rudigoz RC. Birth simulator: reliability of transvaginal assessment of fetal head station as defined by the American College of Obstetricians and Gynecologists classification. Am J Obstet Gynecol. 2005 Mar;192(3):868-74. doi: 10.1016/j.ajog.2004.09.028. PMID 15746684
- [Background] Akmal S, Kametas N, Tsoi E, Hargreaves C, Nicolaides KH. Comparison of transvaginal digital examination with intrapartum sonography to determine fetal head position before instrumental delivery. Ultrasound Obstet Gynecol. 2003 May;21(5):437-40. doi: 10.1002/uog.103. PMID 12768552
- [Background] Ramphul M, Kennelly M, Murphy DJ. Establishing the accuracy and acceptability of abdominal ultrasound to define the foetal head position in the second stage of labour: a validation study. Eur J Obstet Gynecol Reprod Biol. 2012 Sep;164(1):35-9. doi: 10.1016/j.ejogrb.2012.06.001. Epub 2012 Jul 2. PMID 22762840
- [Background] Rozenberg P, Porcher R, Salomon LJ, Boirot F, Morin C, Ville Y. Comparison of the learning curves of digital examination and transabdominal sonography for the determination of fetal head position during labor. Ultrasound Obstet Gynecol. 2008 Mar;31(3):332-7. doi: 10.1002/uog.5267. PMID 18307213
- [Background] Zahalka N, Sadan O, Malinger G, Liberati M, Boaz M, Glezerman M, Rotmensch S. Comparison of transvaginal sonography with digital examination and transabdominal sonography for the determination of fetal head position in the second stage of labor. Am J Obstet Gynecol. 2005 Aug;193(2):381-6. doi: 10.1016/j.ajog.2004.12.011. PMID 16098859
- [Background] Wong GY, Mok YM, Wong SF. Transabdominal ultrasound assessment of the fetal head and the accuracy of vacuum cup application. Int J Gynaecol Obstet. 2007 Aug;98(2):120-3. doi: 10.1016/j.ijgo.2007.05.021. Epub 2007 Jun 22. PMID 17585916